CLINICAL TRIAL: NCT02428387
Title: Evaluation of a Transition Intervention for Family Caregivers of Persons With Alzheimer Disease and Multiple Chronic Conditions
Brief Title: Evaluation of "My Tools 4 Care" for Family Caregivers of Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00048721
Record Dates: First submitted 2015-04-17; First posted 2015-04-28 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Family; Dementia
Keywords: caregivers; intervention; health related quality of life; dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group (Group 1) will receive instructions on how to access "My Tools 4 Care" for 3 months.
  Interventions: Behavioral: My Tools 4 Care
- Educational Control (No Intervention): An educational control group (Group 2) will receive a copy of the Alzheimer's Society' The Progression of Alzheimer's Disease - Overview Booklet.

INTERVENTIONS:
Behavioral: My Tools 4 Care — On-line self-administered (My Tools 4 Care) transition toolkit includes interactive activities and resources to help caregivers deal with their transitions
  Arms: Intervention

SUMMARY:
With the number of Canadians with Alzheimer's disease and related dementias (ADRD) growing, supporting family care partners of persons with ADRD is critical. Family caregivers provide about 90 per cent of in-home care for persons with ADRD, and the care is often difficult due to co-morbidities in persons with ADRD. Family caregivers of older persons with ADRD and multiple chronic conditions (MCC) experience significant, complex, distressing transitions such as changes to their environment, roles and relationships, physical and mental health, isolation, and taking on new tasks. An online Transition Toolkit (My Tools 4 Care) was developed for family caregivers of persons with ADRD and MCC living at home, to support caregivers through transitions and increase their self-efficacy, hope, and quality of life (QOL).

Through this pragmatic mixed methods randomized controlled trial the investigators expect to find that family caregivers receiving the online My Tools 4 Care Toolkit will show greater improvement in hope, self-efficacy and QOL, at no additional cost from a societal perspective, compared with those in an educational control group. Following baseline data collection 180 participants will be randomly assigned to one of the groups with repeated measures at one, three and six months.

DETAILED DESCRIPTION:
Background: With the escalating numbers of persons with Alzheimer Disease and related dementias (ADRD) in Canada, the Rising Tide report suggests that supporting family care partners of persons with AD is critical. Family caregivers provide about 90% of in-home care for persons with ADRD. The care is often difficult and complex due to co-morbidities in persons with ADRD. Family caregivers of older persons with ADRD and MCC experience significant, complex, distressing transitions such as changes to their environment, roles and relationships, physical and mental health, isolation, and taking on new tasks. A Transition Toolkit was developed for family caregivers of persons with AD living at home initially as a paper copy and since has been developed in an on-line format. The purpose of the Toolkit is to support caregivers through transitions and increase their self-efficacy, hope, and quality of life. Sections include About Me, Common Changes to Expect, Frequently Asked Questions, Resources, and Important Health Information. Data from a pilot study of the Toolkit suggest that it is feasible, acceptable, and may support caregivers through transitions. The on-line version of the Toolkit (My Tools 4 Care) includes interactive activities to help caregivers deal with their transitions and as such will be a novel online intervention. The investigators expect that "My Tools 4 Care" will result in improved caregiver outcomes, compared to an educational control group.

Research Questions: (1) Does a transition intervention (My Tools 4 Care) increase hope, self-efficacy and health related quality of life of caregivers of persons with AD and MCC compared with an educational control group from baseline, one month, 3 and 6 months? (2) What are the costs of use of health services at 3 and 6 months of the transition intervention compared with the control group, from a societal perspective? Methods: The design is a pragmatic, multisite, mixed-methods randomized controlled trial (Quantitative +qualitative) with family caregivers of persons >65 years of age who have ADRD and MCC. Participants will be English-speaking family or friends ≥ 18 years of age who provide physical, emotional, or financial care to persons with ADRD. Family caregivers will be recruited through multiple community associations, newspaper ads, posters, the Alberta Caregivers Association, the Alzheimer Society (AS) of Ontario and Alberta. Participants will be randomly assigned to:1) the on-line Transition toolkit (Group 1) or 2) an educational control group (Group 2) who will receive a copy of the Alzheimer's Society's The Progression of Alzheimer's Disease - Overview Booklet. The intervention group (Group 1) will receive instructions on how to access "My Tools 4 Care" for 3 months. To assess dosage of the intervention, caregivers will be asked to document their use of the intervention using a checklist. For the Educational Control Group (Group 2), the participants will receive a copy of the Booklet. Data for all participants will be collected at baseline, and again at 1 month, 3 and 6 months.

Outcome measures are a) hope [Herth Hope Index (HHI)] b) health related quality of life {Short Form 12 (SF-12v2)]) c) self-efficacy [General Self Efficacy Scale (GSES) which measures ability to deal with adverse situations]; and d) use and costs of health services [Health and Social Services Inventory (HSSUI)]. Trained data collectors will administer the instruments using audio-taped telephone interviews at baseline, 1, 3 and 6 months after the start of the intervention. A sample size of 180 caregivers (45 per group x 2 groups x 2 provinces) will provide 80% power (alpha = 0.05) to detect a mean difference of 2 increases in the HHI, GSES, and SF-12 v2, with a standard deviation of 2.5. At 3 months, all participants in group 1 will be interviewed using open-ended questions to further assess perceived effectiveness and mechanisms of change associated with the intervention.

Time Line: Recruitment and data collection will begin April 1, 2015 for 2 years (March 31, 2017). Analysis and report writing April 1, 2017-March 31, 2018.

Expected Outcomes: The investigators expect that family caregivers receiving the on-line Toolkit will show greater improvement in hope, self-efficacy and quality of life at no additional cost from a societal perspective, compared with those receiving the educational brochure.

Impact: The findings of the study will inform policy and practice as the Toolkit can be easily revised for local contexts and scalable in terms of posting on websites such as the Alzheimer Society.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers of persons >65 years of age who have AD and related dementias (ADRD) and MCC (two or more chronic conditions)
* English-speaking
* Family or friends ≥ 18 years of age who provide physical, emotional, or financial care to persons with ADRD and MCC
* Access and able to use a computer (and have an email address).

Exclusion Criteria:

Family caregivers caring for a person with ADRD and MCC who:

* Has died
* Resides in a Long Term Care Facility (nursing home)
* Is hospitalized and designated as restorative care (Alberta) or alternate level of care (Ontario)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2015-04; Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Health Related Quality of Life at One, Three and Six Months | One, three and six months
  SF 12v2 Mental Component and Physical Component Score

SECONDARY OUTCOMES:
Change from Baseline in Hope at One, Three and Six Months | one, three and six months
  Herth Hope Index
Change from Baseline in General Self Efficacy at One, Three and Six Months | One, three and six months
  General Self-Efficacy Scale

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Duggleby, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Jenny Ploeg, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duggleby W, Swindle J, Peacock S. Self-administered intervention for caregivers of persons with Alzheimer's disease. Clin Nurs Res. 2014 Feb;23(1):20-35. doi: 10.1177/1054773812474299. Epub 2013 Feb 6. PMID 23393291
- [Derived] Duggleby W, Ploeg J, McAiney C, Fisher K, Jovel Ruiz K, Ghosh S, Peacock S, Markle-Reid M, Williams A, Triscott J, Swindle J. A Comparison of Users and Nonusers of a Web-Based Intervention for Carers of Older Persons With Alzheimer Disease and Related Dementias: Mixed Methods Secondary Analysis. J Med Internet Res. 2019 Oct 17;21(10):e14254. doi: 10.2196/14254. PMID 31625947
- [Derived] Markle-Reid M, Ploeg J, Valaitis R, Duggleby W, Fisher K, Fraser K, Ganann R, Griffith LE, Gruneir A, McAiney C, Williams A. Protocol for a program of research from the Aging, Community and Health Research Unit: Promoting optimal aging at home for older adults with multimorbidity. J Comorb. 2018 Jul 31;8(1):2235042X18789508. doi: 10.1177/2235042X18789508. eCollection 2018. PMID 30191144
- [Derived] Duggleby W, Ploeg J, McAiney C, Peacock S, Fisher K, Ghosh S, Markle-Reid M, Swindle J, Williams A, Triscott JA, Forbes D, Jovel Ruiz K. Web-Based Intervention for Family Carers of Persons with Dementia and Multiple Chronic Conditions (My Tools 4 Care): Pragmatic Randomized Controlled Trial. J Med Internet Res. 2018 Jun 29;20(6):e10484. doi: 10.2196/10484. PMID 29959111
- [Derived] Duggleby W, Ploeg J, McAiney C, Fisher K, Swindle J, Chambers T, Ghosh S, Peacock S, Markle-Reid M, Triscott J, Williams A, Forbes D, Pollard L. Study protocol: pragmatic randomized control trial of an internet-based intervention (My tools 4 care) for family carers. BMC Geriatr. 2017 Aug 14;17(1):181. doi: 10.1186/s12877-017-0581-6. PMID 28806917